CLINICAL TRIAL: NCT00437216
Title: Phase 4 Open-Label Multicenter Community-based 4-Wk Trial to Assess Efficacy, Tolerance to Tx & Patient Satisfaction w/ CLOBEX® Spray When Used as Mono- or Add-on Therapy to Existing Systemic/Topical Agents for Tx of Plaque Psoriasis
Brief Title: Efficacy, Tolerance and Satisfaction With CLOBEX® Spray When Used as Monotherapy or Add-on Therapy in Plaque Psoriasis
Status: Completed | Type: Observational
Sponsor: Galderma R&D (Industry)
Responsible Party: Ronald W. Gottschalk, MD / Medical Director, Galderma Laboratories, L.P.
Other Study IDs: US10029
Record Dates: First submitted 2007-02-16; First posted 2007-02-19 (Estimated); Last update posted 2022-07-29 (Actual); Status verified 2008-03

CONDITIONS: Psoriasis
MeSH Terms: conditions — Psoriasis | interventions — Clobetasol

STUDY DESIGN:
Observational Model: Case-Only | Time Perspective: Other
Oversight: Data Monitoring Committee: No

GROUPS / COHORTS (2):
- 1: Monotherapy - Subjects who are not currently being treated with anti-psoriatic medication and start using Clobex®
  Interventions: Drug: Clobetasol Propionate, 0.05%
- 2: Add-on therapy - Subjects who are taking some form of anti-psoriatic medication and add Clobex® treatment
  Interventions: Drug: Clobetasol propionate, 0.05% Spray

INTERVENTIONS:
Drug: Clobetasol Propionate, 0.05% — Apply twice daily for 2 or 4 weeks as monotherapy
  Other Names: Clobex® Spray, 0.05%
  Groups: 1
Drug: Clobetasol propionate, 0.05% Spray — Apply twice daily for 2 or 4 weeks as add-on therapy
  Other Names: Clobex® Spray, 0.05%
  Groups: 2

SUMMARY:
Evaluation of the effectiveness of Clobex® Spray, 0.05% when used as monotherapy or add-on therapy to existing systemic or topical anti-psoriatic agents.

DETAILED DESCRIPTION:
Evaluation of the effectiveness of Clobex® Spray, 0.05% when used as monotherapy or add-on therapy to existing systemic or topical anti-psoriatic agents, as determined by the change in the target plaque severity (TPS) rating between Weeks 0 and 4.

ELIGIBILITY:
Inclusion Criteria:

* Moderate to severe plaque psoriasis between 3% and 20% of Body Surface Area (BSA) with a target plaque severity (TPS) of moderate to severe
* At least 1 target site (not on the palms or soles of the feet) with a TPS rating of moderate to severe and with 1 or more elevated, easily palpable, plaques having well-circumscribed margins, and at least 1 cm in diameter
* History of stable plaque psoriasis of greater than or equal to 3 months

Exclusion Criteria:

* Diagnosis of guttate, generalized pustular, erythrodermic, psoriatic arthritis, or nail psoriasis as the sole or predominant form of psoriasis
* Psoriatic arthritis that was not stable or might have required a change in medication during the 4-week study period
* Plaque psoriasis requiring treatment on the face, scalp, neck, groin, and armpits

Ages: 18 Years to 80 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: Community Sample
Sampling Method: Non-Probability Sample
Enrollment: 2488 (Actual)
Dates: Start 2006-02; Primary Completion 2006-07 (Actual); Study Completion 2006-07 (Actual)

PRIMARY OUTCOMES:
Efficacy - Change in Target Plaque Severity rating | 4 weeks

SECONDARY OUTCOMES:
Efficacy - Self-Assessment of Quality of Life, Subject satisfaction | 4 weeks
Safety - Evaluation of adverse events and tolerability | 4 weeks

CONTACTS AND LOCATIONS:
Overall Officials: Ronald W Gottschalk, MD, Study Director — Galderma Laboratories, LP
Locations (1):
- DHC Dimensional HealthCare, Inc. (Clinical Research Organization), Cedar Knolls, New Jersey, United States